CLINICAL TRIAL: NCT03815422
Title: Analgesia Quality and Quality of Deambulation of the Plantar Compartment Block After Hallux Valgus Ambulatory Surgery.
Brief Title: Plantar Compartment Block in Hallux Valgus Ambulatory Surgery
Acronym: Observationnal
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0143
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hallux Valgus Ambulatory Surgery
Keywords: Early ambulation; Plantar block
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Regional anesthesia — Short lasting sciatic nerve block and long lasting plantar block with distal deep peroneal block

SUMMARY:
Hallux valgus surgery is known as a painful surgery. Qualitative pain management is the key to successful early recovery and rehabilitation.

Popliteal sciatic nerve block is widely used despite the risk of falling due to prolonged motor blockade.

Plantar block combined with distal peroneal block may be a better analgesic option in order to provide fast track rehabilitation.

The purpose of this study is to describe the analgesic effect of the plantar compartment block following hallux valgus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* patient covered by social health insurance
* have signed written informed consent
* scheduled for hallux valgus ambulatory surgery

Exclusion Criteria:

* protected patients or patients incapable of giving written informed consent
* pregnant or breastfeeding woman
* vulnerable adult
* inability to participate in pain scoring scales
* severe coagulopathy
* allergy or contraindications to study drugs
* preopérative gait disorders
* chronic kidney disease with glomerular filtration rate (GFR) ≤ 50 ml/min (estimated by the Cockroft and Gault formula)
* severe chronic liver disease
* chronic pain (treated by non steroidal anti inflammatory drugs, opioids, neuroleptic drugs, antidepressant or anticonvulsants)
* peripheral neuropathy
* intervention under general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Plantar compartment block in Hallux Valgus ambulatory surgery
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Analgesia quality of the plantar compartment block | 48 hours
  after Hallux Valgus ambulatory surgery

SECONDARY OUTCOMES:
Quality of deambulation | Quality of deambulation during the first 2 postoperative days.
  48 hours
postoperative analgesic | postoperative analgesic requirement, during the first 2 postoperative days.
  48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fabien SWISSER, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Herteleer M, Choquet O, Swisser F, Bernard N, Gasc A, Canovas F, Dagneaux L, Bringuier S, Capdevila X. Plantar compartment block for hallux valgus surgery: a proof-of-concept anatomic and clinical study. Reg Anesth Pain Med. 2024 Feb 19:rapm-2023-105246. doi: 10.1136/rapm-2023-105246. Online ahead of print. PMID 38373818